CLINICAL TRIAL: NCT04739150
Title: Medical Need Program With Ofev® (Nintedanib) for the Treatment of Adult Patients With Non-IPF (Idiopathic Pulmonary Fibrosis) Chronic Fibrosing Interstitial Lung Diseases (ILDs) With a Progressive Phenotype (PF-ILD's)
Brief Title: An Expanded Access Program in Belgium to Provide Nintedanib to People With Lung Diseases Called Non-IPF ILDs Who Have no Alternative Treatment Options
Status: No longer available | Type: Expanded Access
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1199-0447
Record Dates: First submitted 2021-02-01; First posted 2021-02-04 (Actual); Last update posted 2022-09-09 (Actual); Status verified 2022-09

CONDITIONS: Lung Diseases, Interstitial
MeSH Terms: conditions — Lung Diseases, Interstitial | interventions — nintedanib

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: nintedanib — nintedanib
  Other Names: Ofev®

SUMMARY:
This Expanded Access Program in Belgium is open to people with different lung diseases. This program provides a medicine called nintedanib to people who have no alternative treatment options. They can participate if they have a type of lung disease called non-IPF ILDs (chronic fibrosing interstitial lung diseases with a progressive phenotype other than idiopathic pulmonary fibrosis).

Participants take 2 capsules of nintedanib a day. The treating physician checks the health of the participants and notes health problems that could have been caused by nintedanib. Participants receive nintedanib as long as they benefit or until nintedanib becomes commercially available in Belgium.

For a patient to participate in this program, their treating physician should apply to Boehringer Ingelheim.

ELIGIBILITY:
Inclusion Criteria:

* The patient is not eligible for a clinical trial running with Ofev® and/or a clinical trial running in the envisaged indication of this program.
* The patient cannot be satisfactorily treated with the approved and commercially available alternative treatments, in accordance with clinical guidelines, because of efficacy and/or safety issues.
* Signed informed consent form
* Age ≥ 18 years
* Patients diagnosed with ILD who fulfilled at least 1 of the following criteria for PF-ILD within 24 months prior to inclusion in this Medical Need Program (MNP):

  * Clinically significant decline in Forced Vital Capacity (FVC) % predicted based on a relative decline of ≥10%
  * Marginal decline in FVC % predicted based on a relative decline of ≥5 to <10% combined with worsening of respiratory symptoms
  * Marginal decline in FVC % predicted based on a relative decline of ≥5% to <10% combined with increasing extent of fibrotic changes on chest high resolution computed tomography (HR-CT) imaging
  * Worsening of respiratory symptoms as well as increasing extent of fibrotic changes on chest HR-CT imaging.
* The treating physician must be a qualified pulmonologist with sufficient experience in treating patients with ILD and sufficient knowledge to administer Ofev®, and states to comply with the following requirements to claim this experience:

  * Participates/has participated in clinical trials, in the scope of interstitial lung diseases or has fulfilled a residency or fellowship program in ILD
  * Is part of a multidisciplinary team, that has treated ≥25 ILD patients within a random uninterrupted timeframe of 24 months
  * The multidisciplinary team exists at least of the following specialist physicians with experience in management of interstitial lung diseases: a pulmonologist, a radiologist, a pathologist, and a rheumatologist.

Exclusion Criteria:

* The safety, efficacy, and pharmacokinetics of nintedanib have not been studied in patients with severe renal impairment (<30 ml/min creatinine clearance). These patients are therefore excluded from the program.
* The safety and efficacy of nintedanib have not been investigated in patients with hepatic impairment classified as Child Pugh B and C. Treatment of patients with moderate (Child Pugh B) and severe (Child Pugh C) hepatic impairment with Ofev® is not recommended.
* The safety and efficacy of Ofev® in children aged 0-18 years have not been established. No data are available. Non-adult patients are therefore excluded.
* Hypersensitivity to nintedanib, to peanut or soya, or to any of the excipients listed in section 6.1. of the SMPC.
* Diagnosis of IPF as Ofev® can be obtained through reimbursed product in this indication.
* Patients at known risk for bleeding including patients with inherited predisposition to bleeding or patients receiving a full dose of anticoagulative treatment were not included in the clinical trials. Non-serious and serious bleeding events, some of which were fatal, have been reported in the post-marketing period (including patients with or without anticoagulant therapy or other medicinal products that could cause bleeding). Therefore, these patients should only be treated with Ofev if the anticipated benefit outweighs the potential risk.
* Ofev® should not be used in patients with severe pulmonary hypertension.
* Patients with a recent history of myocardial infarction or stroke. Further exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (14):
- Belgium (14):
  - Aalst - HOSP Onze-Lieve-Vrouw, Aalst
  - ULB Hopital Erasme, Anderlecht
  - Ziekenhuis Netwerk Antwerpen (ZNA) - Campus Middelheim, Antwerp
  - AZ Klina, Brasschaat
  - Universitair Ziekenhuis Brussel, Brussels
  - Brussels - UNIV Saint-Luc, Brussels
  - UNIV UZ Gent, Ghent
  - Jessa Ziekenhuis - Campus Virga Jesse, Hasselt
  - Kortrijk - HOSP AZ Groeninge Kennedylaan, Kortrijk
  - UZ Leuven, Leuven
  - Centre Hospitalier Universitaire de Liège, Liège
  - Roeselare - HOSP AZ Delta, Roeselare
  - Sint-Niklaas - HOSP AZ Nikolaas (Campus St-Niklaas), Sint-Niklaas
  - Yvoir - UNIV UCL de Mont-Godinne, Yvoir

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com